CLINICAL TRIAL: NCT06896786
Title: Sodium Management Tool in Hemodialysis Patients
Brief Title: This Study Evaluates the Impact of the Sodium Management Tool (SMT) on Hemodialysis Patient Outcomes Compared to Standard Care
Acronym: SOMEDIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sharon-Rose Maloney (Other)
Responsible Party: Sponsor-Investigator, Sharon-Rose Maloney, MD, Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEP-LU-0001
Record Dates: First submitted 2025-02-09; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hemodialysis; Interdialytic Weight Gain; Intradialytic Hypotension
Keywords: sodium management in hemodialyis patients; management of complaints in hemodialysis patients; interdialytic weight gain; intradialytic hypotension; sodium management tool

STUDY DESIGN:
Intervention Model Description: randomised, cross over , single site design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): dialysis conducted with standard of care
- dialysis assisted with the sodium management tool (Active Comparator): dialysis assisted with the sodium management tool
  Interventions: Other: dialysis assisted with the sodium management tool

INTERVENTIONS:
Other: dialysis assisted with the sodium management tool — Sodium management tool is a modul of the fresenius 6008 dialysis machine. This model approximates changes in plasma electrolyte concentrations during dialysis and allows the estimation of sodium concentration based on dialysate conductivity. Na control biosensor continuously (every minute) monitors the dialysate side sodium balance based on measurements of fresh and spent dialysate conductivities and the application of a kinetic model to account for the typical influence of other ions on dialysate conductivity. In activated Na control, as "zero diffusive" mode, dialysate sodium is then adjusted continuously to minimize diffusive Na transfer. SMT is part of the 6008 Machine and its certification is included in the Fresenius 6008 Machine certification. Untill now there is no data if this modul benefits. in this study the investigator compares standard of care dialysis (Arm 1) with dialysis assisted with the SMT (Arm ) on clinical outcome
  Arms: dialysis assisted with the sodium management tool

SUMMARY:
Title of the Study: Sodium Management Tool in Hemodialysis Patients

Brief Summary:

The goal of this clinical trial is to learn whether the Sodium Management Tool (SMT) can improve patients clnical outcomes.

The main questions this study aims to answer are:

Does the SMT help reduce weight gain between dialysis sessions? Does the SMT improve dialysis tolerance by reducing symptoms like low blood pressure and muscle cramps?

Researchers will compare standard dialysis to dialysis using the SMT to see if clinical outcomes are better in dialysis that use the SMT.

Participants will:

Receive dialysis three times per week with either standard dialysis or SMT-activated dialysis Switch between standard dialysis and SMT-activated dialysis after 4 weeks Have their blood pressure, sodium levels, and symptoms monitored during treatment Report their symptoms and thirst levels in a questionnaire Some participants may continue for an additional 4 weeks with a personalized SMT setting based on their symptoms and weight changes.

This study will help determine whether the SMT can improve sodium balance and make dialysis more comfortable for patients.

DETAILED DESCRIPTION:
Title of the Study: Sodium Management Tool in Hemodialysis Patients

Objectives This study aims to evaluate the impact of the Sodium Management Tool (SMT) by Fresenius on interdialytic weight gain and dialysis tolerance in hemodialysis patients. While the SMT is already in use across various dialysis centers, there is currently no systematic data collection regarding its clinical benefits.

In conventional hemodialysis, a fixed dialysate sodium concentration (typically 136-138 mmol/L) is used without adjustments during dialysis. If the dialysate sodium concentration is higher than the plasma sodium level, sodium can diffuse into the patient, leading to increased thirst and interdialytic weight gain. These factors are associated with higher mortality and an increased risk of cardiovascular events. Conversely, a negative sodium balance (dialysate sodium concentration lower than plasma sodium) can reduce plasma tonicity, increasing the risk of muscle cramps and intradialytic hypotension.

The SMT continuously measures plasma sodium concentration (once per minute) and adjusts the dialysate sodium concentration. This optimization of sodium homeostasis may reduce the occurrence of muscle cramps and hypotensive episodes during dialysis.

Methods The study will include all outpatient hemodialysis patients from the Lucerne Cantonal Hospital at the Luzern, Luzern Süd, and Sursee sites who undergo dialysis three times per week with Fresenius 6008 machines and have provided informed consent.

Participants will be randomized into two groups:

Group 1: Standard dialysis procedure in weeks 1-4, followed by dialysis with the SMT activated in weeks 5-8. The SMT will be set to 0 mmol/L, meaning the dialysate sodium concentration will be adjusted so that the plasma sodium level at the end of dialysis matches the pre-dialysis level.

Group 2: Dialysis with the SMT activated (Na 0 mmol/L) in weeks 1-4, followed by standard dialysis in weeks 5-8.

Data collection includes:

Interdialytic weight gain Pre- and post-dialysis plasma sodium levels Blood pressure before and after dialysis Bolus administration and total sodium removal Symptomatic hypotension, blood pressure drops >20 mmHg, and muscle cramps (documented by nursing staff) Dialysis tolerance and thirst perception, assessed using a visual analog scale (VAS) Patient-reported symptoms (thirst, shortness of breath, muscle cramps, dizziness, fatigue) using the Dialysis Symptom Index Extension Phase (Weeks 9-12)

For a subset of participants, the study will continue:

Subgroup A: Patients with high interdialytic weight gain will have the SMT set to -1 mmol/L. This setting aims for a plasma sodium level 1 mmol/L lower at the end of dialysis, enhancing sodium removal.

Subgroup B: Patients frequently experiencing symptoms (cramps, hypotension) will have the SMT set to +1 mmol/L. This adjustment targets a plasma sodium level 1 mmol/L higher at the end of dialysis, increasing plasma tonicity.

Outcomes Primary Outcome: Effect of the SMT on interdialytic weight gain. Secondary Outcomes: Incidence of intradialytic hypotension, muscle cramps, and specific patient symptoms (thirst, fatigue, shortness of breath, muscle cramps) measured using the Dialysis Symptom Index.

The study will be conducted in accordance with the Declaration of Helsinki and the International Conference on Harmonization (ICH-GCP) guidelines for Good Clinical Practice. All participants will provide written informed consent. Confidentiality and data protection will be maintained at all times.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients on hemodialysis for at least three months,
* Dialysis three times a week, age >/= 18,
* dialysis with a Fresenius 6008 Machine,
* signed informed consent

Exclusion:

* Dialysis access with repeated Interruption due to flow problems
* plasma natrium < 130 mmol/l, > 145 mmol/l, pregnancy -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
mean relative interdialytic weight gain (rIDWG) | measured in the last week of each study period (week 4 ,8 ,12)
  The primary endpoint is the mean relative interdialytic weight gain (rIDWG) measured in the last week of each study period. Interdialytic weight gain (IDWGt): Weight measured at the beginning of the dialysis at time t minus weight measured after the dialysis at time t-1 (weight pre-dialysis t - weight post-dialysis t-1)
  Relative interdialytic weight gain (rIDWGt)): Difference of the weight measured at the beginning of the dialysis at time t and the weight measured after the dialysis at time t-1, divided by the weight measured after the dialysis at time t-1 ((weight pre-dialysis t - weight postdialysis t-1) / weight post-dialysis t-1)

SECONDARY OUTCOMES:
dialysis tolerance with and without SMT based on dialysis symptom index (DSI) | measured in the last week of each study period (week 4, 8 and 12)
  To assess dialysis tolerance with and without SMT based on PROMs:
  specific sodium/volume related complaints from the dialysis symptom index (DSI): dry mouth , muscle cramps , dizziness, tiredness , shortness of breath ,VAS Dialysis tolerance , VAS Thirst intensity
  DSI: For each question, the presence or absence of a specific symptom, as well as its severity, is assessed using a five-point Likert scale, with each response ranging from 0 to 4 (i.e., a response of "0" indicates "no," whereas a response of "4" indicates "yes: very much")
dialysis tolerance with and without SMT based on Visual Analogue Scale (VAS ) Dialysis tolerance: | measured in the last week of each study period (week 4, 8 and 12)
  To assess dialysis tolerance with and without SMT based on VAS for Dialysis tolerance
  VAS Dialyse tolerance: Patients will be requested to rate their dialysis experience on a 10-cm VAS, where 0 is the worst imaginable dialysis experience and 10 the best imaginable dialysis experience.
Thirst Intensity with and without SMT based on VAS thirst intensity | measured in the last week of each study period (week 4, 8 and 12)
  To assess thirst intensity with and without SMT based on VAS for thirst intensity
  VAS thirst intensity: Patients will be requested to rate their thirst since the last dialysis on a 10-cm VAS, with 0 indicating no thirst and 10 indicating the worst possible thirst.

CONTACTS AND LOCATIONS:
Overall Officials: Balthasar Hug, Professor, Principal Investigator — LUKS Luzern

IPD SHARING:
Plan to Share IPD: No